CLINICAL TRIAL: NCT00002862
Title: A PHASE I STUDY OF PERILLYL ALCOHOL IN PATIENTS WITH REFRACTORY MALIGNANCIES (NSC #641066)
Brief Title: Perillyl Alcohol in Treating Patients With Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065133; YALE-HIC-8895; NCI-T96-0064D
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2000-09

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — perillyl alcohol

ARMS (1):
- Arm I (Experimental): Groups of 3-6 patients receive escalating doses of oral perillyl alcohol three times per day until the maximum tolerated dose or recommended phase II dose is determined. Treatment at the assigned dose continues until disease progression or unacceptable toxicity intervenes. Patients with stable disease after 8 weeks of treatment are removed from study.
  Interventions: Drug: perillyl alcohol

INTERVENTIONS:
Drug: perillyl alcohol

SUMMARY:
Phase I trial to study the effectiveness of perillyl alcohol in treating patients with refractory cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Estimate the maximum tolerated dose of perillyl alcohol given chronically three times per day in patients with refractory malignancies.

II. Describe the toxic effects and pharmacokinetics associated with this regimen.

III. Evaluate any antitumor activity of perillyl alcohol in these patients. IV. Assess the ability of perillyl alcohol to induce tumor differentiation and reduce telomerase activity in patients from whom serial biopsies can be obtained.

OUTLINE: This is a dose escalation study to determine the maximum tolerated dose of perillyl alcohol.

Groups of 3-6 patients receive escalating doses of oral perillyl alcohol three times per day until the maximum tolerated dose or recommended phase II dose is determined. Treatment at the assigned dose continues until disease progression or unacceptable toxicity intervenes. Patients with stable disease after 8 weeks of treatment are removed from study.

Patients are followed for duration of response and survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid malignancy or lymphoma for which no effective therapy exists
* Measurable or evaluable disease
* No CNS metastasis unless stable for at least 4 weeks following surgery and/or radiotherapy and no requirement for anticonvulsants

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-2
* Life expectancy: At least 3 months
* ANC at least 1,500
* Platelets at least 100,000
* Bilirubin no greater than 2.0 mg/dL
* AST less than 2.5 times normal
* Creatinine clearance at least 50 mL/min
* No concurrent cholesterol-lowering agents
* No active infection (including HIV)
* No concomitant medical condition that precludes study compliance
* No pregnant or nursing women
* Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since chemotherapy (6 weeks since nitrosoureas or mitomycin)
* At least 4 weeks since wide-field radiotherapy
* Fully recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1996-10; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Murren, MD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States